CLINICAL TRIAL: NCT06982313
Title: Long-term Follow-up of the TAM-01 Study, a Phase III Trial of Low Dose Tamoxifen in Breast DCIS and Premalignant Disease
Brief Title: Long-term Follow-up of the TAM-01 Study
Acronym: TAM-01 L_FU
Status: Not yet recruiting | Type: Observational
Sponsor: Ente Ospedaliero Ospedali Galliera (Other)
Responsible Party: Principal Investigator, Andrea DeCensi, Dr., Ente Ospedaliero Ospedali Galliera
Other Study IDs: TAM-01 long-term follow-up
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer Invasive
Keywords: Low-Doses; Breast Cancer; Tamoxifen; Long-term follow up; DCIS; clinical trial, phase III; breast intraepithelial neoplasia; precancerous conditions; biomarkers; Insulin-Like Growth Factor Binding Proteins
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Precancerous Conditions | interventions — Tamoxifen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Tamoxifen: All women received one tablet of tamoxifen 5 mg per day for 3 years during the TAM-01 phase III trial.
  Interventions: Drug: Tamoxifen (Nolvadex)
- Placebo: All women received one tablet of placebo per day for 3 years during the TAM-01 phase III trial.
  Interventions: Drug: Tamoxifen (Nolvadex) placebo

INTERVENTIONS:
Drug: Tamoxifen (Nolvadex) — 5 mg per day for 3 years during TAM-01 phase III trial
  Groups: Tamoxifen
Drug: Tamoxifen (Nolvadex) placebo — Tamoxifen (Nolvadex) placebo per day for 3 years during TAM-01 phase III trial.
  Groups: Placebo

SUMMARY:
Low-dose tamoxifen (5 mg/day for three years, BabyTam) has emerged as a safer and effective alternative to the standard regimen (20 mg/day), reducing breast cancer recurrence with fewer adverse events. The TAM-01 phase III trial demonstrated a 42% reduction in breast cancer events over ten years compared to placebo in women with ductal carcinoma in situ (DCIS) or high-risk lesions (HRL, ADH, LCIS), supporting its inclusion in clinical guidelines.

The phase III TAM-01 trial enrolled 500 women, comparing low-dose tamoxifen to placebo over three years, with a median follow-up of 9.7 years (IQR, 8.3-10.9). Results showed a significant reduction in invasive breast cancer (HR = 0.58; 95% CI: 0.35-0.95; p = 0.03) and in contralateral breast cancer, CBC (HR = 0.36; 95% CI: 0.14-0.92; p = 0.025), with no increase in serious adverse events.

Exploratory analyses suggested a greater benefit in postmenopausal women (HR = 0.30; 95% CI: 0.11-0.82), compared to premenopausal women (HR = 0.73; 95% CI: 0.30-1.76), though this interaction did not reach statistical significance (p-interaction = 0.13). However, our unpublished data indicate a remarkable reduction of CBC in premenopausal women on BabyTam.

The TAM-01 long-term follow-up study aims to extend the follow-up of TAM-01 participants, evaluating long-term outcomes, including incidence of invasive breast cancer and DCIS, with a focus on tumor laterality and menopausal status as well as to assess other non-invasive events (LCIS, ADH or ALH) and adverse outcomes of special interest.

The findings are expected to strengthen the evidence supporting low-dose tamoxifen as a viable prevention strategy in high-risk populations with intraepithelial neoplasia (IEN or DCIS+HRLs).

DETAILED DESCRIPTION:
Low-dose tamoxifen (5 mg/day for three years) has emerged as a safer alternative to standard-dose tamoxifen (20 mg/day), effectively reducing the risk of breast cancer recurrence while minimizing adverse events. The TAM-01 phase III trial demonstrated that this regimen decreased subsequent breast cancer events by 42% compared to placebo after 10 years in women with ductal carcinoma in situ (DCIS) or high-risk lesions (atypical ductal hyperplasia, ADH, or lobular carcinoma in situ, LCIS), without exceeding serious adverse events and patient-reported outcomes, thus supporting its wide uptake in the medical community and NCCN guideline inclusion.

The IBIS-I trial reinforced the role of tamoxifen in breast cancer prevention, demonstrating a lasting reduction in breast cancer incidence, particularly in estrogen receptor-positive tumors, with benefits extending beyond the treatment period. Furthermore, real-world evidence indicates strong patient preference for low-dose tamoxifen due to its reduced side effects, increasing adherence in clinical practice. Additionally, studies have shown that low-dose tamoxifen can lower mammographic density, potentially improving screening sensitivity and facilitating earlier cancer detection.

The TAM-01 (EudraCT number: 2007-007740-10) trial was a multicenter, phase III trial comparing 5 mg/day tamoxifen to placebo over 3 years in 500 women aged 75 years or younger with an ECOG performance status of 1 or lower, and hormone-sensitive (ER or progesterone receptor ≥ 1%) or unknown DCIS (69%) or breast intraepithelial neoplasia (ADH, 20% or LCIS, 11%). Women with high-grade or comedo/necrotic DCIS were treated with adjuvant radiotherapy at 50 Gy in 25 fractions. Participants were followed up every 6 months, undergoing annual mammography and transvaginal ultrasound for 3 years of treatment and then being seen annually for 7 years of follow-up. All breast-related events during the trial were centrally adjudicated by an expert committee. The primary endpoint was the incidence of invasive breast cancer and DCIS.

The mean (SD) age at treatment initiation was 54 (9) years, with 58% being postmenopausal women. After a median follow-up of 9.7 years (IQR, 8.3 to 10.9 years), 66 breast cancers were diagnosed (15 in situ; 51 invasive): 25 in the tamoxifen group and 41 in the placebo group (annual rate per 1,000 person-years: 11.3 with tamoxifen vs. 19.5 with placebo; hazard ratio [HR] 0.58; 95% CI, 0.35 to 0.95; p = 0.03). The majority of recurrences were invasive (77%) and ipsilateral (59%). For contralateral breast cancer incidence, there were 6 events in the tamoxifen group and 16 in the placebo group (HR, 0.36; 95% CI, 0.14 to 0.92; p = 0.025). No differences were observed between the groups regarding patient-reported outcomes (menopausal symptoms) or serious adverse events during the extended follow-up period.

An exploratory analysis from TAM-01 suggested that the efficacy of low-dose tamoxifen may differ by menopausal status. Although a protective effect was observed in both groups, the reduction appeared more pronounced in postmenopausal women (HR: 0.30; 95% CI, 0.11 to 0.82) than in premenopausal women (HR: 0.73; 95% CI, 0.30 to 1.76). Although this difference did not reach statistical significance (p-interaction = 0.13), it raises important questions about the biological mechanisms underlying tamoxifen's effects and the role of estradiol levels in modulating its efficacy.

The importance of identifying the optimal dose of tamoxifen is underscored by studies demonstrating that lower doses can retain efficacy while significantly reducing adverse effects, supporting the integration of low-dose regimens into prevention strategies. Randomized trials, such as those by Eriksson et al. and Bhatia et al., have shown the potential of low-dose tamoxifen in diverse populations, including high-risk individuals and those with preinvasive breast cancer.

Recent findings from a preplanned biomarker analysis of the TAM-01 trial have provided further support for the role of low-dose tamoxifen in targeted breast cancer prevention strategies. Specifically, baseline levels of insulin-like growth factor binding protein-3 (IGFBP-3) in the top three quartiles (≥3.44 μg/mL), but not in the lowest quartile, were shown to predict greater efficacy of BabyTam compared with placebo (p-interaction = 0.006). In contrast, baseline levels of IGF-I, estradiol, or sex hormone-binding globulin (SHBG) were not predictive of BabyTam efficacy, whereas the IGF-I/IGFBP-3 molar ratio showed a borderline significant interaction (p-interaction = 0.067). This study unveils the potential of serum biomarkers, specifically IGFBP-3 and IGF-I/IGFBP-3 ratios, as predictive factors of BabyTam efficacy among individuals with DCIS or high-risk lesions. These findings hold significant implications in clinical practice, offering a means to discern patients who may derive maximal benefits from BabyTam.

The previous TAM-01 study discontinued the follow-up of enrolled patients because, under Regulation (EU) No 536/2014 on clinical trials on medicinal products for human use, the study would have had to be migrated to the Clinical Trials Information System (CTIS) managed by the European Medicines Agency (EMA).

As the study had started in 2008, both the protocol and the entire study documentation were not compliant with the requirements of the Regulation (EU) No 536/2014. For both administrative and feasibility reasons, the migration was not possible, and the original study was therefore closed and replaced by the current version.

Based on the TAM-01 findings, this long-term follow-up study aims to compare the long-term outcomes in women who participated in the TAM-01 trial. By extending the follow-up, the study aims to compare the incidence of invasive breast cancer and DCIS, considering tumor laterality and menopausal status, as well as to assess other non-invasive events (LCIS, ADH or ALH) and adverse outcomes of special interest.

The results of this study are expected to provide a robust evidence base for the incorporation of low-dose tamoxifen into routine clinical practice and to address personalized preventive strategies in high-risk populations.

ELIGIBILITY:
Inclusion criteria:

* Women previously enrolled in the TAM-01 trial (EudraCT number: 2007-007740-10).
* Written informed consent.

Exclusion criteria:

* None.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all women previously enrolled in the TAM-01 study (EudraCT number: 2007-007740-10).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2035-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of invasive breast cancer and ductal carcinoma in situ (DCIS) | Each patient will be followed for a total period of 20 years from the date of randomization in the TAM-01 trial, with data collected and updated annually.
  The primary objective is to compare the incidence of invasive breast cancer and ductal carcinoma in situ in a long-term follow-up of the TAM-01 study.
Incidence of invasive breast cancer and ductal carcinoma in situ (DCIS) considering tumor laterality and menopausal status | Each patient will be followed for a total period of 20 years from the date of randomization in the TAM-01 trial, with data collected and updated annually.
  To compare the incidence of invasive breast cancer and DCIS by tumor site (ipsilateral or contralateral) and menopausal status.

SECONDARY OUTCOMES:
Incidence of other non-invasive events | Each patient will be followed for a total period of 20 years from the date of randomization in the TAM-01 trial, with data collected and updated annually.
  The incidence of other non-invasive events, such as lobular carcinoma in situ (LCIS), atypical ductal hyperplasia (ADH) or atypical lobular hyperplasia (ALH).
Overall Survival and Breast Cancer Survival (OS) | Each patient will be followed for a total period of 20 years from the date of randomization in the TAM-01 trial, with data collected and updated annually.
  Overall Survival and Breast Cancer Survival (OS)
Adverse Events | Each patient will be followed for a total period of 20 years from the date of randomization in the TAM-01 trial, with data collected and updated annually.
  The incidence of adverse events, including endometrial cancer, deep vein thrombosis or pulmonary embolism, other neoplasms, coronary heart disease, bone fracture and cataract. These events will be expressed as the number of events and percentage (%) within each treatment arm, allowing for a direct comparison between the two groups.
Biomarkers evaluation | Each patient will be followed for a total period of 20 years from the date of randomization in the TAM-01 trial, with data collected and updated annually.
  Association between biomarker levels (particularly IGFBP-3) and clinical outcomes, aimed at assessing their prognostic and/or predictive value in the context of long-term follow-up.

OTHER OUTCOMES:
Exploratory Endpoint: Correlation between biomarkers | Each patient will be followed for a total period of 20 years from the date of randomization in the TAM-01 trial, with data collected and updated annually
  Correlation between biomarkers collected at baseline, at year one, at the end of treatment and two years after treatment completion and long-term clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Censi, MD, Principal Investigator — E. O. Ospedali Galliera
Locations (1):
- E. O. Ospedali Galliera, Genoa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: TAM-01 study (EudraCT number: 2007-007740-10). — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2007-007740-10
- See also: TAM-01 study (ClinicalTrials.gov ID: NCT01357772). — https://www.clinicaltrials.gov/study/NCT01357772